CLINICAL TRIAL: NCT02930941
Title: Topical Intranasal Tranexamic Acid for Epistaxis in the Emergency Department
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminate due to slow enrollment rate.
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 844609
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Results first posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Epistaxis
Keywords: tranexamic acid; epistaxis; emergency medicine; intranasal; TXA
MeSH Terms: conditions — Epistaxis | interventions — Tranexamic Acid; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Tranexamic Acid (100 mg/mL) (Experimental): TXA (100 mg/1mL) sprayed in to the affected nostril(s) via intranasal atomization device. May repeat 2 doses in each affected nostril(s).
  Interventions: Drug: Tranexamic Acid
- 0.9% Sodium Chloride (Placebo Comparator): 0.9% Sodium Chloride (1mL) in to the affected nostril(s) via intranasal atomization device. May repeat 2 doses in each affected nostril(s).
  Interventions: Drug: 0.9% Sodium Chloride

INTERVENTIONS:
Drug: Tranexamic Acid — TXA (100 mg/1mL) in to the affected nostril(s) via intranasal atomization device. May repeat 2 doses in each affected nostril(s).
  Other Names: Cyklokapron
  Arms: Tranexamic Acid (100 mg/mL)
Drug: 0.9% Sodium Chloride — 0.9% Sodium Chloride (1mL) in to the affected nostril(s) via intranasal atomization device. May repeat 2 doses in each affected nostril(s).
  Other Names: Saline solution
  Arms: 0.9% Sodium Chloride

SUMMARY:
It is estimated that epistaxis results in 4.5 million emergency department visits per year throughout the United States. Due to the adverse effects of standard treatment options for epistaxis, tranexamic acid (TXA) may be considered an attractive option. In previous studies, when used with nasal packing, TXA showed faster time to control of bleeding. The goal of this study is to determine the efficacy and safety of topical intranasal TXA applied via atomizer for patients with epistaxis who present to the emergency department.

DETAILED DESCRIPTION:
This is a prospective, randomized, single-center, double-blinded, placebo controlled study comparing efficacy and safety of topical intranasal tranexamic acid for epistaxis. The primary outcome was time to control of bleeding and secondary outcomes were length of stay in the emergency department, re-bleeding within the first 24 hours, and re-bleeding at one week. Safety outcomes were the incidence of thromboembolic events and other drug-related adverse events.

Patients aged 18 years of age or older and diagnosed with anterior epistaxis were included. Patients were excluded if they were unable to consent, do not have a valid telephone number, pregnant women, prisoners, cognitively impaired individuals, diagnosis of posterior epistaxis, major trauma, bleeding disorder (such as thrombocytopenia or hemophilia), hemodynamically unstable, or had a known hypersensitivity to study medication.

Patients were randomly assigned to tranexamic acid treatment group or placebo group. After consenting, patients received TXA (100 mg/1mL) or 0.9% sodium chloride (1 mL) in to the affected nostril(s) via intranasal atomization device. If bleeding did not cease, two repeat doses were allowed and after twenty minutes of continued bleeding the study physician could treat with any additional treatment options. Patients were contacted via telephone within one week to inquire about incidences of re-bleeding or any complications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with anterior epistaxis

Exclusion Criteria:

* Unable to consent, do not have a valid telephone number, pregnant women, prisoners, cognitively impaired individuals, diagnosis of posterior epistaxis, major trauma, bleeding disorder (such as thrombocytopenia or hemophilia), hemodynamically unstable, or had a known hypersensitivity to study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-02; Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Moulin, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morgan DJ, Kellerman R. Epistaxis: evaluation and treatment. Prim Care. 2014 Mar;41(1):63-73. doi: 10.1016/j.pop.2013.10.007. PMID 24439881
- [Background] Dunn CJ, Goa KL. Tranexamic acid: a review of its use in surgery and other indications. Drugs. 1999 Jun;57(6):1005-32. doi: 10.2165/00003495-199957060-00017. PMID 10400410
- [Background] Pallin DJ, Chng YM, McKay MP, Emond JA, Pelletier AJ, Camargo CA Jr. Epidemiology of epistaxis in US emergency departments, 1992 to 2001. Ann Emerg Med. 2005 Jul;46(1):77-81. doi: 10.1016/j.annemergmed.2004.12.014. PMID 15988431
- [Background] Kucik CJ, Clenney T. Management of epistaxis. Am Fam Physician. 2005 Jan 15;71(2):305-11. PMID 15686301
- [Background] Villwock JA, Jones K. Recent trends in epistaxis management in the United States: 2008-2010. JAMA Otolaryngol Head Neck Surg. 2013 Dec;139(12):1279-84. doi: 10.1001/jamaoto.2013.5220. PMID 24136624
- [Background] Singer AJ, Blanda M, Cronin K, LoGiudice-Khwaja M, Gulla J, Bradshaw J, Katz A. Comparison of nasal tampons for the treatment of epistaxis in the emergency department: a randomized controlled trial. Ann Emerg Med. 2005 Feb;45(2):134-9. doi: 10.1016/j.annemergmed.2004.10.002. PMID 15671968
- [Background] White A, O'Reilly BF. Oral tranexamic acid in the management of epistaxis. Clin Otolaryngol Allied Sci. 1988 Feb;13(1):11-6. doi: 10.1111/j.1365-2273.1988.tb00275.x. PMID 3286068
- [Background] Tibbelin A, Aust R, Bende M, Holgersson M, Petruson B, Rundcrantz H, Alander U. Effect of local tranexamic acid gel in the treatment of epistaxis. ORL J Otorhinolaryngol Relat Spec. 1995 Jul-Aug;57(4):207-9. doi: 10.1159/000276741. PMID 7478455
- [Background] Zahed R, Moharamzadeh P, Alizadeharasi S, Ghasemi A, Saeedi M. A new and rapid method for epistaxis treatment using injectable form of tranexamic acid topically: a randomized controlled trial. Am J Emerg Med. 2013 Sep;31(9):1389-92. doi: 10.1016/j.ajem.2013.06.043. Epub 2013 Jul 30. PMID 23911102
- [Background] Utkewicz MD, Brunetti L, Awad NI. Epistaxis complicated by rivaroxaban managed with topical tranexamic acid. Am J Emerg Med. 2015 Sep;33(9):1329.e5-7. doi: 10.1016/j.ajem.2015.02.049. Epub 2015 Mar 6. No abstract available. PMID 25895714
- [Background] Klepfish A, Berrebi A, Schattner A. Intranasal tranexamic acid treatment for severe epistaxis in hereditary hemorrhagic telangiectasia. Arch Intern Med. 2001 Mar 12;161(5):767. doi: 10.1001/archinte.161.5.767. No abstract available. PMID 11231712
- [Background] Aguilera X, Martinez-Zapata MJ, Hinarejos P, Jordan M, Leal J, Gonzalez JC, Monllau JC, Celaya F, Rodriguez-Arias A, Fernandez JA, Pelfort X, Puig-Verdie Ll. Topical and intravenous tranexamic acid reduce blood loss compared to routine hemostasis in total knee arthroplasty: a multicenter, randomized, controlled trial. Arch Orthop Trauma Surg. 2015 Jul;135(7):1017-25. doi: 10.1007/s00402-015-2232-8. Epub 2015 May 7. PMID 25944156
- [Background] Waldow T, Szlapka M, Haferkorn M, Burger L, Plotze K, Matschke K. Prospective clinical trial on dosage optimizing of tranexamic acid in non-emergency cardiac surgery procedures. Clin Hemorheol Microcirc. 2013 Jan 1;55(4):457-68. doi: 10.3233/CH-131782. PMID 24113504
- [Background] Wolfe TR, Braude DA. Intranasal medication delivery for children: a brief review and update. Pediatrics. 2010 Sep;126(3):532-7. doi: 10.1542/peds.2010-0616. Epub 2010 Aug 9. PMID 20696726
- [Background] Reuben A, Appelboam A, Stevens KN, Vickery J, Ewings P, Ingram W, Jeffery AN, Body R, Hilton M, Coppell J, Wainman B, Barton A. The Use of Tranexamic Acid to Reduce the Need for Nasal Packing in Epistaxis (NoPAC): Randomized Controlled Trial. Ann Emerg Med. 2021 Jun;77(6):631-640. doi: 10.1016/j.annemergmed.2020.12.013. Epub 2021 Feb 19. PMID 33612282
- [Background] Akkan S, Corbacioglu SK, Aytar H, Emektar E, Dagar S, Cevik Y. Evaluating Effectiveness of Nasal Compression With Tranexamic Acid Compared With Simple Nasal Compression and Merocel Packing: A Randomized Controlled Trial. Ann Emerg Med. 2019 Jul;74(1):72-78. doi: 10.1016/j.annemergmed.2019.03.030. Epub 2019 May 9. PMID 31080025

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tranexamic Acid (100 mg/mL) | 0.9% Sodium Chloride
Started | 17 | 18
Completed | 16 | 16
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- TXA Group: Patients that received tranexamic (TXA)(100 mg/1mL) sprayed in to the affected nostril(s) via intranasal atomization device. May repeat 2 doses in each affected nostril(s).
- NS Group: Patients that received 0.9% Sodium Chloride (NS) (1mL) in to the affected nostril(s) via intranasal atomization device. May repeat 2 doses in each affected nostril(s).
- Total: Total of all reporting groups
Arm/Group | TXA Group | NS Group | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 10 | 9 | 19
Age, Continuous [Mean (Full Range); unit: years] | 61 [28 to 83] | 62 [21 to 95] | 62 [21 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 18
  Male | 11 | 6 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 35
Past Medical History [Count of Participants; unit: Participants]
  Anemia | 1 | 1 | 2
  Atrial Fbrillation or flutter | 4 | 2 | 6
  Cancer | 2 | 2 | 4
  Chronic Kidney Disease | 5 | 2 | 7
  Congestive Heart Failure | 4 | 1 | 5
  Diabetes | 4 | 6 | 10
  Hyperlipidemia | 5 | 5 | 10
  Ischemic Stroke | 1 | 0 | 1
  Obesity | 2 | 0 | 2
  Pulmonary Embolism | 0 | 1 | 1
  Deep Vein Thrombosis | 0 | 1 | 1
  Myocardial infarction | 1 | 0 | 1
  Coronary Artery Bypass | 1 | 1 | 2
  Hypertension | 11 | 7 | 18
Antiplatelet [Count of Participants; unit: Participants]
  Aspirin | 8 | 2 | 10
  Clopidogrel | 2 | 1 | 3
  Prasugrel | 1 | 0 | 1
  Ticagrelor | 1 | 0 | 1
Anticoagulation [Count of Participants; unit: Participants]
  Warfarin | 4 | 2 | 6
  Apixaban | 3 | 2 | 5
  Rivaroxaban | 0 | 0 | 0
  Dabigatran | 0 | 0 | 0
Hemoglobin [Mean (Full Range); unit: g/dL] — grams (g) per decilitre (dL)
  g/dL | 12.9 [8.2 to 15.4] | 12 [7.5 to 15.7] | 12.4 [7.5 to 15.7]
Hematocrit [Mean (Full Range); unit: % by volume of hemoglobin in blood] — percentage by volume of hemoglobin in blood
  % by volume of hemoglobin in blood | 38 [25.7 to 45] | 35.8 [23.2 to 45.6] | 36.9 [23.2 to 45.6]
Platelet [Mean (Full Range); unit: x10^3 per microliter] — x10^3 per microliter
  x10^3 per microliter | 210.1 [103 to 300] | 248 [122 to 419] | 229.8 [103 to 419]

OUTCOME MEASURES:

1. Primary Outcome: Time to Control of Bleeding (Minutes, Median, Interquartile Range)
Description: Time to control of bleeding was defined as the time from the start of enrollment and direct pressure and administration of study drug to the resolution of bleeding
Time Frame: During emergency department (ED) visit
Population: Intention-to-treat
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- TXA Group: Tranexamic (TXA)(100 mg/1mL) sprayed in to the affected nostril(s) via intranasal atomization device. May repeat 2 doses in each affected nostril(s).
- NS Group: 0.9% Sodium Chloride (NS) (1mL) in to the affected nostril(s) via intranasal atomization device. May repeat 2 doses in each affected nostril(s).
Arm/Group | TXA Group | NS Group
Number analyzed (Participants) | 17 | 18
minutes | 64 [33 to 104] | 42 [26 to 131]

2. Secondary Outcome: Length of Stay in the Emergency Department (Minutes, Median, Inter-Quartile Range)
Description: Length of stay was defined as time from enrollment in study to discharge from the emergency department
Time Frame: During emergency department (ED) visit
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | TXA Group | NS Group
Number analyzed (Participants) | 17 | 18
minutes | 268 [195 to 607] | 346 [283 to 410]

3. Secondary Outcome: Number of Participants With Re-bleeding at 24 Hours
Description: The number of participants with re-bleeding at 24 Hours was evaluated during follow up phone call
Time Frame: 24 hours
Population: Intention to treat. Lost to follow up: 1 in TXA group and 1 in NS group
Measure: Count of Participants; unit: Participants
Groups:
- TXA Group: Tranexamic group
- NS Group: Normal saline
Arm/Group | TXA Group | NS Group
Number analyzed (Participants) | 16 | 17
Participants | 3 | 9

4. Secondary Outcome: Number of Participants With Re-bleeding at One Week
Description: The number of participants with re-bleeding at one week was evaluated during the follow-up phone call
Time Frame: 7 days
Population: Intention-to-treat. Loss to follow-up: 1 in TXA group and 2 in NS group
Measure: Count of Participants; unit: Participants
Arm/Group | TXA Group | NS Group
Number analyzed (Participants) | 16 | 16
Participants | 2 | 6

5. Secondary Outcome: Thromboembolism
Description: Patient reported thromboembolic events during follow-up phone calls at 24 hours and at one week
Time Frame: 7 days
Population: Intention to treat. Lost to follow up of 1 in TXA group and 2 in NS group.
Measure: Count of Participants; unit: Participants
Arm/Group | TXA Group | NS Group
Number analyzed (Participants) | 16 | 16
Participants | 0 | 0

6. Secondary Outcome: Drug-Related Adverse Events
Description: Patient-reported drug-related adverse events during ED visit
Time Frame: during emergency department (ED) visit
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | TXA Group | NS Group
Number analyzed (Participants) | 17 | 18
Participants
  Nasal burning | 2 | 0
  Nasal irritation | 0 | 0
  Unpleasant taste | 1 | 0

ADVERSE EVENTS:
Time Frame: One week from initial ED visit
Description: All adverse effects reported from patients were collected. Mortality was not collected beyond 7 days.
Arm/Group | TXA Group | NS Group
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 4/17 | 0/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TXA Group (N=17) | NS Group (N=18)
Nasal Burning (General disorders) | 2 (2) | 0 (0)
Unpleasant taste (General disorders) | 1 (1) | 0 (0)
Rhinorrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Coronavirus Disease 2019 (COVID-19) pandemic significantly impacted the ability to enroll patients; early termination leading to a small number of patients; single-center study;

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2017-02-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT02930941/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2017-02-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT02930941/SAP_001.pdf